CLINICAL TRIAL: NCT02488304
Title: Prospective Study for Transplant Optimization Using Functional Imaging (TROFI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the lung transplantation program at the site is on hold
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUI-2015-141
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2017-10

CONDITIONS: Bronchiolitis Obliterans; Lung Transplant Rejection
Keywords: HRCT; High Resolution Computed Tomography scans; Functional Respiratory Imaging; FRI; Computed Tomography; CT; Bronchiolitis Obliterans Syndrome; BOS; Lung Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HRCT scans (Experimental): High Resolution Computed Tomography scans will be taken
  Interventions: Radiation: HRCT scans

INTERVENTIONS:
Radiation: HRCT scans — A HRCT scan at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC) will be taken on visit 2, visit 3, visit 4, visit 5, visit 6, and visit 7.
  An upper airway (UA) scan will be taken on visit 2.
  Other Names: High Resolution Computed Tomography scans

SUMMARY:
The objective of this study is to detect BOS in an early stage by using the outcome parameters generated by Functional Respiratory Imaging (FRI). Robust and automated segmentation algorithms will be developed for these parameters, focusing on quantitative computed tomography (CT) image analyses to provide the physician a more sensitive diagnostics tool. The evolution of rejection over time will be monitored using non-rigid image registration methods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years old
* Written informed consent obtained
* Patients who are planned to receive a lung transplant in the near future
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before screening visit and will continue to use a contraception method during the study
* The patient must be able to perform the lung monitoring at home

Exclusion Criteria:

* Pregnant or lactating female
* Known history of or active airways or anastomotic complications requiring intervention such as stenting or dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Airway Volume (iVaw) using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Airway Resistance (iRaw) using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7. Airway resistance is defined as the pressure drop over the airways divided by the airflow.
Change in Specific Airway Volume (siVaw) using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Specific Airway Resistance (siRaw) using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Lobe Volumes (iVlobes) using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Air trapping using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7. Air trapping is defined as the regions in the lung with a gray value on the CT-scan image smaller than -850 HU at functional residual capacity.
Change in Internal Lobar Airflow Distribution using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7. Airflow distribution is defined in as the percentage of air going to every lobe when inhaling from FRC to TLC and is calculated for every lobe as: IALDlobe [%] = 100 (VTLC_lobe - VFRC_lobe) / (VTLC_lungs - VFRC_lungs).
Change in Low Attenuation or Emphysema Score using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Blood Vessel Density or Fibrosis Score using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.
Change in Airway Wall Thickness using FRI | 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months post-transplant
  Exploratory imaging endpoints: HRCT scan will be taken at visit 2- visit 7.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, M.D., M.S., Principal Investigator — University Hospital of Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium